CLINICAL TRIAL: NCT01472900
Title: A Randomized Split-Face Controlled Trial Comparing Efficacy of 2940 Nanometer Er:YAG Laser to 2.5% BP Gel for the Treatment of Inflammatory Acne
Brief Title: 2940nm Er:YAG Laser Versus Benzoyl Peroxide Gel for the Treatment of Inflammatory Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattaporn Rojarayanont, M.D., Faculty of Medicine, Department of Medicine, Dermatological unit, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERYAG-AC01
Record Dates: First submitted 2011-11-12; First posted 2011-11-17 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Solid-State; clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Er:YAG laser (Experimental)
  Interventions: Device: 2940 nm Er:YAG laser (DualisXS M002-2A, Fotona®, Fotona d.d, Ljubljana, Slovenia)
- BP gel (Active Comparator)
  Interventions: Drug: Benzoyl Peroxide gel

INTERVENTIONS:
Device: 2940 nm Er:YAG laser (DualisXS M002-2A, Fotona®, Fotona d.d, Ljubljana, Slovenia) — 2 passes of 2940nm Er:YAG laser
  Other Names: DualisXS M002-2A, Fotona®, Fotona d.d, Ljubljana, Slovenia
  Arms: Er:YAG laser
Drug: Benzoyl Peroxide gel — 2.5% benzoyl peroxide gel apply twice daily on inflammatory acne on the control side of face
  Other Names: 2.5% benzoyl peroxide gel
  Arms: BP gel

SUMMARY:
Acne is one of the most common conditions that patients seek for help in dermatological clinic. Nowadays, conventional treatment including topical agents(retinoids, antibiotics ,antiseptics and keratolytic agents) and systemic agents( antibiotics and retinoids) give a satisfying result but not to every patient. Some patients are not well respond to conventional therapy while some patients are unable to tolerate side effects of the treatments. Therefore, interventions to reduce acne are vigorously experimented . Lights and lasers including intense pulsed light, pulsed dye laser with or without photosensitizer and infrared lasers have been found to be useful in treating active inflammatory acne. Although,pain ,downtime and poor response of comedonal acne are limitations of those lights and lasers therapy. 2940 nm Erbium:YAG laser which has both resurfacing and photothermal effects is our laser of interest to seek for its efficacy in the treatment of inflammatory acne.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year-old to 45 year-old
* Mild to moderate severity of acne vulgaris with at least 5 active inflammatory acne lesions on each side of the face and less than 25% difference in lesion count between each side of face
* Fitzpatrick skin phototype I-IV

Exclusion Criteria:

* History or clinical presentation of hypertrophic scar or keloid
* Photoaggravated skin diseases i.e. systemic lupus erythematosus, polymorphous light eruption, solar urticaria
* Oral isotretinoin taken within the last 6 months prior to enrollment
* Topical retinoid within 4 weeks prior to enrollment
* Systemic acne therapies (oral antibiotics) within 4 week prior to enrollment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
percentage change from baseline of inflammatory acne lesion count at 6 week after 1st 2940nm Er:YAG laser treatment | 6 week
  % change from baseline = (NV- NB)/NB x 100% NV = number of lesion at each visit NB = number of lesion at baseline

SECONDARY OUTCOMES:
Safety | week0,2,4
  Safety profile of 2940nm Er:YAG laser for the treatment of inflammatory acne including;
  * Visual analogue scale of pain score
  * Adverse events(AEs) include types of AEs(erythema, pain/burning sensation, dryness/excessive scaling, pigmentary change), timing, intenstity, outcome and action taking regarding to study procedure particular subject.
Photographic clinical improvement | week 2,4,6 and 10
  Photographic clinical improvement of acne, acne scar, erythema, hyperpigmentation and overall improvement by blinded dermatologists using quartile grading system comparing baseline and each clinical visit (week 2,4,6 and 10)
Patient satisfaction | week 6
  Self evaluation of patient satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- See also: Management of acne: a report from a Global Alliance to Improve Outcomes in Acne — http://www.ncbi.nlm.nih.gov/pubmed/12833004
- See also: Persistent acne in women : implications for the patient and for therapy — http://www.ncbi.nlm.nih.gov/pubmed/17007539
- See also: The quality of life in acne: a comparison with general medical conditions using generic questionnaires — http://www.ncbi.nlm.nih.gov/pubmed/10233319
- See also: New insights into the management of acne: an update from the Global Alliance to Improve Outcomes in Acne group — http://www.ncbi.nlm.nih.gov/pubmed/19376456
- See also: Prevalence and severity of facial and truncal acne in a referral cohort — http://www.ncbi.nlm.nih.gov/pubmed/18561586
- See also: Profile of acne vulgaris--a hospital-based study from South India — http://www.ncbi.nlm.nih.gov/pubmed/19439880
- See also: Guidelines of care for acne vulgaris management — http://www.ncbi.nlm.nih.gov/pubmed/17276540